CLINICAL TRIAL: NCT00312975
Title: Phase 2 Randomized, Non-Comparative Study Of CP-675,206 Or Best Supportive Care Immediately Following First-Line, Platinum-Based Therapy In Patients With Stage IIIB (With Effusion) Or Stage IV Non-Small Cell Lung Cancer That Has Responded Or Remained Stable
Brief Title: Randomized Study Of CP-675,206 or Best Supportive Care Immediately After Platinum-Based Therapy For Non-Small Cell Lung Cancer (NSCLC)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: A3671015
Record Dates: First submitted 2006-04-07; First posted 2006-04-11 (Estimated); Last update posted 2012-06-07 (Estimated); Status verified 2012-06

CONDITIONS: Carcinoma, Non-small-cell Lung
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — tremelimumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm A (Experimental)
  Interventions: Drug: CP-675,206
- Arm B (Active Comparator)
  Interventions: Drug: best supportive care

INTERVENTIONS:
Drug: CP-675,206 — Given intravenously every 3 months
  Arms: Arm A
Drug: best supportive care — As per investigator discretion. Excludes chemotherapy or other anti-cancer therapy
  Arms: Arm B

SUMMARY:
The purpose of this trial is to study how long patients can remain progression free when they receive CP-675,206, compared to how long patients can remain progression free when they receive best supportive care. If you choose to take part, you will be randomized to receive either CP-675,206 as maintenance therapy or best supportive care. Best supportive care means you will not receive any study drug or other treatment for your cancer. Best supportive care could include treatment with antibiotics, analgesic drugs (medicine for pain), blood transfusions or psychosocial and nutritional support, depending on your needs. You have a 50% chance of being randomized to receive CP-675,206.

ELIGIBILITY:
Inclusion Criteria:

* Stage IIIb (with effusion) or stage IV disease that has responded or remained stable after 6 cycles of a platinum containing 1st-line regimen
* Patients must be able to be randomized between 3 and no more than 6 weeks after the last dose of first-line therapy.

Exclusion Criteria:

* No other systemic therapy except 1st-line platinum based treatment
* Symptomatic or uncontrolled brain mets or uncontrolled pleural effusions.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2006-05; Primary Completion 2008-04 (Actual); Study Completion 2010-02 (Actual)

PRIMARY OUTCOMES:
The length of time until there is evidence of disease progression in patients treated with CP-675,206 and in patients receiving best supportive care. | 3 months to 2 years from randomization

SECONDARY OUTCOMES:
Survival | 2 years
Levels of study drug in blood samples taken at specified time points. | up to 2 years
Whether polymorphisms of certain genes influence safety. | up to 2 years
Health-related quality of life outcomes. | up to 2 years
Tumor response | up to 2 years
Number of patients with adverse events as a measure of safety of CP-675,206 when administered to patients with NSCLC | up to 2 years
Blood levels of any human anti-human antibody response | up to 2 years
Immune response. | up to 2 years
Efficacy | up to 2 years

CONTACTS AND LOCATIONS:
Locations (22):
- United States (13):
  - Research Site, Bentonville, Arkansas
  - Research Site, Fayetteville, Arkansas
  - Research Site, Orange, California
  - Research Site, Danbury, Connecticut
  - Research Site, Atlanta, Georgia
  - Research Site, Lexington, Kentucky
  - Research Site, Alexandria, Louisiana
  - Research Site, New York, New York
  - Research Site, Oneida, New York
  - Research Site, Oswego, New York
  - Research Site, Syracuse, New York
  - Research Site, Canton, Ohio
  - Research Site, Philadelphia, Pennsylvania
- Canada (3):
  - Research Site, Calgary, Alberta
  - Research Site, Edmonton, Alberta
  - Research Site, Montreal, Quebec
- Czechia (3):
  - Research Site, Prague
  - Research Site, Tábor
  - Research Site, Ústí nad Labem
- Research Site, Seoul, South Korea
- United Kingdom (2):
  - Research Site, Southampton, Hampshire
  - Research Site, London